CLINICAL TRIAL: NCT01334229
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Effects of Sitagliptin on the Kinetics of Triglyceride-rich Lipoproteins Apolipoprotein B48 and Apolipoprotein B100 in Patients With Type 2 Diabetes
Brief Title: Sitagliptin and Kinetics of Triglyceride-rich Lipoproteins Apolipoprotein B48 and B100 in Patients With Type 2 Diabetes
Acronym: JANUB48
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patrick Couture, MD, PhD, FRCP, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIS#39262
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: sitagliptin; diabetes; apolipoprotein B48 and B100
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg/d for 6 weeks
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg/d for 6 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Placebo for 6 weeks
  Arms: Placebo

SUMMARY:
Sitagliptin is a potent and selective inhibitor of dipeptidyl peptidase IV (DPP-IV), and has been shown to reduce fasting and postprandial glucose levels in patients with type 2 diabetes mainly through incretin hormone-mediated improvements in islet function [13]. Although clinical studies to date indicate that fasting lipid levels are minimally affected by DPP-IV inhibitor treatment [14-16], animal studies suggested that DPP-IV inhibition reduce intestinal triglycerides (TG) absorption and apolipoprotein (apo) production [17] and increased chylomicron catabolism [18]. Interestingly, a recent study supporting this hypothesis showed that vildagliptin therapy was able to reduce postprandial intestinal triglyceride-rich lipoproteins (TRL) particles in patients with type 2 diabetes [19]. Recently, our group has reported that sitagliptin treatment significantly reduced plasma apo B-48 and TG concentrations in the postprandial state. Moreover, animal studies showed that sitagliptin decreased intestinal secretion of intestinal apo B-48, mainly by increasing level of glucagon-like peptide (GLP)-1 [20]. Therefore, the present study was designed to examine the effects of sitagliptin on the kinetics of TRL apo B-48 and in patients with type 2 diabetes. A possible reduction in postprandial atherogenic TRL apo B-48-containing lipoprotein levels by sitagliptin would add to therapeutic utility of this DPP-4 inhibitor and suggest the potential to reduce cardiovascular risk in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 65 years of age.
* Post-menopausal women under age 65 on stable medical therapy for 6 months before the study (the patient should have demonstrated stable lipid panels)
* Women should not be on hormone replacement therapy (no recent starting or stopping)
* Type 2 diabetes as defined by the American Diabetes Association.
* Non-smoker.
* Body mass index between 25.0 and 40.0 kg/m2.
* Baseline glycated hemoglobin A1c (HbA1c) between 6.5 and 8.5%.
* Baseline fasting plasma glucose < 15.0 mmol/L.
* Plasma triglyceride levels between 1.5 and 8.0 mmol/L (135 and 710 mg/dl) at screening and week -4.
* Patients having received stable doses of metformin for at least 3 months before randomization.
* Subjects must be willing to give written informed consent and able to adhere to dosing schedule, visit schedule and phone follow-up assessment.
* Patients should be otherwise generally healthy, without elevations in hepatic transaminases or abnormal renal function or coagulation.
* Patients having normal thyroid stimulating hormone at screening

Exclusion Criteria:

* Patients with extreme dyslipidemias, such as familial hypercholesterolemia will be excluded.
* Patients with type 1 diabetes, secondary form of diabetes or acute metabolic diabetic complications will be excluded.
* Patients having received or being treated with insulin or a thiazolidinedione within the past 6 months will be excluded.
* Patients taking any other hypoglycemic agent, other than metformin.
* Subjects will be excluded if they have cardiovascular disease (coronary heart disease, cerebrovascular disease or peripheral arterial disease) or if they are taking other medications known to affect lipoprotein metabolism (e.g. steroids, beta blockers, thiazide diuretics, lipid lowering agents, significant alcohol intake etc.).
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Individuals with a history of mental instability, drug or alcohol abuse or individuals who have been treated or are being treated for severe psychiatric illness that, in the opinion of the investigator, may interfere with optimal participation in the study.
* History of alcohol or drug abuse within the past 2 years. Patients must not take alcohol during the study.
* Disorders of the hematologic, digestive, or central nervous systems, including cerebrovascular disease and degenerative disease, that would limit study evaluation or participation.
* Known impairment of renal function (serum creatinine levels > 1.7 mg/dL for men), dysproteinemia, nephrotic syndrome, or other renal disease (24-hour urinary protein ≥3 ± 1 g).
* Active or chronic hepatobiliary or hepatic disease. In addition, patients with aspartate aminotransferase or alanine aminotransferase >2 x upper limit of the laboratory reference range will be excluded.
* Subjects with coagulopathy (prothrombin time or partial thromboplastin time at Visit 1 >1.5 times control).
* Subjects with hemoglobin >2 x the lower limit of the laboratory reference range will be excluded.
* Patients who are known to have tested positive for human immunodeficiency virus (HIV).
* Patients who are currently enrolled in another clinical study.
* Patients who have used any investigational drug within 30 days of the first clinic visit.
* Congestive heart failure New York Heart Association (NYHA) Class III or IV. Uncontrolled cardiac arrhythmias within 3 months of study entry.
* Uncontrolled diabetes mellitus (HbA1c>8.5%) or other endocrine or metabolic disease known to influence serum lipids or lipoproteins. Clinically euthyroid subjects on replacement doses of thyroid hormone are eligible for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin Then Placebo: First intervention: Sitagliptin 100 mg/d for 6 weeks Washout: 4 weeks Second intervention: Placebo for 6 weeks
- Placebo First Then Sitagliptin: First intervention: Placebo for 6 weeks Washout: 4 weeks Second intervention: Sitagliptin 100 mg/d for 6 weeks
Period: Overall Study
Arm/Group | Sitagliptin Then Placebo | Placebo First Then Sitagliptin
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin First Then Placebo: First intervention: Sitagliptin 100 mg/d for 6 weeks Washout: 4 weeks Second intervention: Pacebo for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Sitagliptin First Then Placebo | Placebo First Then Sitagliptin | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (4.6) | 59 (2.9) | 58.2 (3.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Apolipoprotein B48 and Apolipoprotein B100 Production Rates With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 22 | 22
mg/kg/day
  apolipoprotein B48 production rate | 2.1 (0.7) | 2.5 (1.2)
  apolipoprotein B100 production rate | 27.5 (8.4) | 30.3 (11.3)

2. Secondary Outcome: Measurement of Glucagon-like Peptide-1 by ELISA
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 22 | 22
pmol/L | 5.6 (6.8) | 3.1 (5.8)

3. Secondary Outcome: Measurement of Glucose
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 22 | 22
mmol/L | 7.7 (1.2) | 8.9 (1.5)

4. Secondary Outcome: Measurement of Insulin
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 22 | 22
pmol/L | 161.1 (91.7) | 179.5 (88.1)

5. Secondary Outcome: Measurement of Apolipoprotein B48 and Apolipoprotein B100 Pool Sizes With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 22 | 22
mg
  apolipoprotein B48 pool size | 38.4 (25.8) | 48.5 (45.2)
  apolipoprotein B100 pool size | 488.0 (210.2) | 537.8 (232.0)

6. Secondary Outcome: Measurement of Apolipoprotein B48 and Apolipoprotein B100 Fractional Catabolic Rates With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pools/day
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 22 | 22
pools/day
  apolipoprotein B48 fractional catabolic rate | 6.2 (2.5) | 6.3 (3.2)
  apolipoprotein B100 fractional catabolic rate | 5.9 (2.3) | 5.9 (2.6)

ADVERSE EVENTS:
Arm/Group | Placebo | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No